CLINICAL TRIAL: NCT05044702
Title: Effects of Retro Walking on Pain, Physical Function and Flexibility in Chronic Non-specific Low Back Pain
Brief Title: Effects of Retro Walking in Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/0126
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retro walking (Experimental): Retro walking
  Interventions: Other: Retro walking; Other: conventional physical therapy
- conventional physical therapy (Active Comparator): Conventional Physical therapy
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: Retro walking — Retro walking will be performed on treadmill for 15 min per day for 3 days per week for 4 weeks at self-paced speed.
  Arms: Retro walking
Other: conventional physical therapy — hot pack for 10 mints and conventional exercise program Conventional physiotherapeutic exercise program which consist of exercises such as
  * prone leg extension
  * prone lying chest elevation
  * prone extension with alternate arm and leg lift
  * supine bridging, bridging with one leg lift Each exercise will be performed as 2 sets of 12 repetitions of each exercise, each exercise position maintained for 10 s, and a rest of 1 min between the sets will be perform. No external load/resistance will be provided for the exercises, and the participants will be perform the exercise within their available range of motion

SUMMARY:
Chronic low back pain (CLBP) is a clinical entity that can be defined as back pain with duration of more than 12 weeks. Chronic low back pain is associated with restriction in daily physical activities that ultimately leads to disuse atrophy of muscles. Moreover, weak and atrophied muscles around the lumbar spine cause immense immobility and recurring low back pain in these patients. The objective of this study will be to determine the effect of retro walking on pain, physical function and flexibility in chronic non-specific low back pain.

This study will be a randomized controlled trial and will be conducted in physiotherapy department in DHQ hospital Nankana Sahib. The study will be completed in time duration of six months after the approval of synopsis and consecutive sampling technique will be used. 40 subjects will be divided in two groups. Group A will follow retro walking and conventional treatment while group B will follow only conventional treatment. Data will be collected by all participants before 1st session after 6th session and at the end of 12th session by using NPRS, MODI, sit and reach test and Modified schobber's test. Data will be analyzed by SPSS-25.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a clinical entity that can be defined as back pain with duration of more than 12 weeks. Epidemiologic evidence suggests that 50% of the general population experiences CLBP and around 70% have encountered at least one occurrence of it during their lifetime.Chronic low back pain is associated with restriction in daily physical activities that ultimately leads to disuse atrophy of muscles.Moreover, weak and atrophied muscles around the lumbar spine cause immense immobility and recurring low back pain in these patients The prevalence of low back pain increases peak between 35-55 years of age.Low back pain is caused by a degenerated or damaged facet joint or sacroiliac joint with soft tissue injury on the trunk or by lumbar instability from weakened muscle strength.Lumbar instability restricts muscle strength, endurance, flexibility, and active range of motion (AROM). In particular, patients with Chronic low back pain (CLBP) persisting for more than 6 months restrict trunk movement to minimize pain in the lumbosacral area or leg, which aggravates the level of lumbar muscle weakness in paraspinal muscles and the multifidus.These changes increase lumbar instability and raise the recurrence of low back pain. Patients with CLBP suffer from deteriorated physical functions and production activities due to weakened muscle strength in the lumbar region.

In 2015 Yun Ha Park et al, conducted a study to confirm the effect of various forms of walking on health related physical fitness, lumbar muscle strength, range of motion and the pain index. Forty females were divided into 4 groups: walking forward (n=10), walking backward (n=10), walking forward & backward (n=10), and control group (n=10). All participants in walking groups walked 50 min/day and 3 days/week during 10 weeks. The results of study concluded that walking forward, walking backward, and walking forward & backward caused significant changes in health related physical fitness, lumbar muscle strength, ROM and pain. Especially the group of walking backward showed low figures in pain.

In a study conducted by Kim SH et al, in 2016 twenty five unilateral exercise athlete were included. The purpose of this study was to investigate the effect of backward walking on isokinetic muscular function, low back pain index and lumbo sacral angle in unilateral exercise athletes. Backward walking was performed with a frequency of three times a week by 60 minutes at a time for 10 weeks. Comparison of related variables before and after backward walking was verified. This study concluded that backward walking improves muscle strength of the lumbar vertebra and reduces the lumbosacral angle and appeared to reduce the pain of the lumbar vertebra.

In an experimental study conducted by Manisha Rathi et al in 2017, 30 women having mechanical low back pain were divided in 2 groups Group A and Group B. Group A underwent core strengthening exercises and hot pack for 10 min, and Group B underwent same protocol along with Retro-walking for 10 min, the protocol was given for 4 weeks, outcome measures were NPRS at rest and activity and core strength. Results showed that there was significant reduction in NPRS at rest and activity in both the groups but group B showed more reduction.

In 2018 Ansari B et al, conducted an experimental study to investigate the electromyographic activity of lumbar multifidus (MF) and erector spinae (ES) muscle during forward walking (FW) and backward walking (BW) in participants with and without chronic low back pain (CLBP). 25 health and 25 chronic low back pain patients was included. Study concluded that BW leads to greater activation of the paraspinal muscles. Along with global extensor (ES), activity of core extensor (MF) is also higher during BW than FW in both healthy participants and CLBP patients. BW is a more favorable aerobic activity to enhance lumbar para spinal recruitment. These findings may have important clinical implications in the rehabilitation of CLBP.

In a study conducted by Ansari S et al, in 2020 thirty athletes with low back pain were randomly assigned in two groups. One group was given conventional treatment and other was given retro walking and conventional treatment. . Pain, flexion range of motion, balance, and muscle fatigability were examined before and after 4 weeks of the intervention. Study concluded that retro walking when added to conventional exercises may be helpful in reducing chronic mechanical LBP and improving dynamic balance but has no additional effect in improving the flexion range of motion and reducing muscle fatigability.

The literature has proved the significant effects of retro walking on pain, balance, and range of motion in athletes, but its effects on physical function, pain and flexibility of hamstrings and flexibility of lumbar spine in chronic non- specific low back pain in general population are still needed to be investigated further. The objective of current study will be to determine the effects of retro walking on pain, physical function and flexibility in chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age:25-45yrs
* LBP for>12 weeks
* those having mild-to-moderate disability
* An ODI score ranging from 20 to 60%
* Being able to walk independently with or without walking aids
* Being able to understand and follow instructions on testing procedures.

Exclusion Criteria:

* Any recent trauma leading to body pain and postural deformities
* Any previous surgery leading to body pain and postural deformities,
* congenital postural deformities,
* current pregnancy,
* Nerve root compression (determined by the presence of two or more of the symptoms-weakness of myotomes, sensory loss of dermatomes, and hyporefexia),
* sacroiliac joint dysfunction (determined by any three positives among distraction test, gaenslen's test, thigh thrust test, sacral thrust test, and compression test),
* any metabolic or vascular disease with a neurological component such as atherosclerosis
* Any contraindication to physiotherapy

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
• Numeric Pain Rating Scale (NPRS) | 4 weeks
  NPRS is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
MODIFIED OSWESTRY LOW BACK DISABILITY QUESTIONNAIRE | 4 weeks
  The MODI has been developed to assess pain related disability. The questionnaire consists of 10 items addressing different aspects of function. Each item is scored from 0 to 5, with higher values representing greater disability. The total score is multiplied by 2 and expressed as a percentage

SECONDARY OUTCOMES:
MODIFIED SCHOBER TEST | 4 weeks
  It is commonly used assessment methods for lumbar flexion ROM. To perform this test, the examiner puts his thumbs on the inferior margin of the subject's PSIS. An ink mark is drawn along the midline of the lumbar spine horizontal to the PSIS (lower landmark). While the examiner holds the tape firmly against the subject's skin, he marks a second line 15 cm above the original one (higher landmark). Then the subject is asked to do an active anterior flexion of the trunk without increasing the pain. The new distance between the lower and higher landmarks is then measured. The subject returns to the neutral position. The difference in the initial distance between the skin markings in the neutral position and the new measurements made in the flexion position is used to indicate the amount of lumbar flexion. Measurements are recorded to the nearest mm
SIT-AND-REACH TEST | 4 weeks
  Sit-and-reach test (SR) are commonly used to evaluate the hamstring and lower back flexibility. The subjects sit with their feet approximately hip-wide against the testing box. They keep their knees extended and place the right hand over the left, and slowly reach forward as far as they could by sliding their hands along the measuring board

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Study Chair — Riphah International University
Locations (1):
- Physical therapy Center in DHQ hospital, Nankana Sahib, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smeets RJ, Wade D, Hidding A, Van Leeuwen PJ, Vlaeyen JW, Knottnerus JA. The association of physical deconditioning and chronic low back pain: a hypothesis-oriented systematic review. Disabil Rehabil. 2006 Jun 15;28(11):673-93. doi: 10.1080/09638280500264782. PMID 16809211
- [Background] Chatzitheodorou D, Kabitsis C, Malliou P, Mougios V. A pilot study of the effects of high-intensity aerobic exercise versus passive interventions on pain, disability, psychological strain, and serum cortisol concentrations in people with chronic low back pain. Phys Ther. 2007 Mar;87(3):304-12. doi: 10.2522/ptj.20060080. Epub 2007 Feb 6. PMID 17284546
- [Background] Hoogkamer W, Meyns P, Duysens J. Steps forward in understanding backward gait: from basic circuits to rehabilitation. Exerc Sport Sci Rev. 2014 Jan;42(1):23-9. doi: 10.1249/JES.0000000000000000. PMID 24188982
- [Background] Viggiano D, Travaglio M, Cacciola G, Di Costanzo A. Effect of backward walking on attention: possible application on ADHD. Transl Med UniSa. 2014 Dec 19;11:48-54. eCollection 2015 Jan-Apr. PMID 25674550
- [Background] Ansari B, Bhati P, Singla D, Nazish N, Hussain ME. Lumbar Muscle Activation Pattern During Forward and Backward Walking in Participants With and Without Chronic Low Back Pain: An Electromyographic Study. J Chiropr Med. 2018 Dec;17(4):217-225. doi: 10.1016/j.jcm.2018.03.008. Epub 2019 Jan 20. PMID 30846913
- [Background] Tousignant M, Poulin L, Marchand S, Viau A, Place C. The Modified-Modified Schober Test for range of motion assessment of lumbar flexion in patients with low back pain: a study of criterion validity, intra- and inter-rater reliability and minimum metrically detectable change. Disabil Rehabil. 2005 May 20;27(10):553-9. doi: 10.1080/09638280400018411. PMID 16019864
- [Background] Lopez-Minarro PA, Andujar PS, Rodrnguez-Garcna PL. A comparison of the sit-and-reach test and the back-saver sit-and-reach test in university students. J Sports Sci Med. 2009 Mar 1;8(1):116-22. eCollection 2009. PMID 24150564